CLINICAL TRIAL: NCT03512210
Title: A Single-arm Study to Evaluate the Feasibility and Efficacy of a Minimal Monitoring Strategy to Deliver Pan-genotypic Ribavirin-free HCV Therapy to HCV Infected Populations Who Are HCV Treatment Naïve With Evidence of Active HCV Infection: The MINMON Study
Brief Title: Monitoring SOF/VEL in Treatment Naïve, HCV Participants With Active Infection
Acronym: MINMON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5360; UM1AI068636 (NIH)
Record Dates: First submitted 2018-04-19; First posted 2018-04-30 (Actual); Results first posted 2021-07-16 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Hepatitis C; HIV-1-infection; Liver Diseases
MeSH Terms: conditions — Hepatitis C; Liver Diseases | interventions — Sofosbuvir; velpatasvir; sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MINMON 24 weeks with SOF/VEL 12 Weeks (Experimental): Participants received Sofosbuvir/Velpatasvir (SOF/VEL [Tradename: Epclusa®]) tablet for 12 weeks with a minimal monitoring (MINMON) strategy for 24 weeks
  Interventions: Drug: Sofosbuvir/Velpatasvir (SOF/VEL); Other: Minimal Monitoring (MINMON) Strategy

INTERVENTIONS:
Drug: Sofosbuvir/Velpatasvir (SOF/VEL) — 400/100 mg fixed-dose combination (FDC) tablet administered orally once daily with or without food.
  Other Names: Epclusa
Other: Minimal Monitoring (MINMON) Strategy — MINMON Strategy:
  1. No pre-treatment HCV genotyping
  2. Entire treatment course (84) tablets of SOF/VEL administered to participants at study entry
  3. No scheduled on-treatment laboratory monitoring or clinic visits
  4. Remote contact with participants at week 4 and week 22

SUMMARY:
To achieve global hepatitis C virus (HCV) elimination by 2030, 80% of the ~71 million people with chronic HCV infection will need to be treated, necessitating simplification of treatment delivery and associated laboratory monitoring without compromising efficacy or safety. The COVID-19 pandemic has further highlighted the need for innovative models of health care delivery that minimize face-to-face patient-provider contact. The purpose of this study was to evaluate the feasibility, safety, and efficacy of a minimal monitoring (MINMON) strategy to deliver interferon- and RBV-free, pan-genotypic DAA therapy to treat active HCV in HCV treatment naïve participants.

DETAILED DESCRIPTION:
This study evaluated the feasibility, safety, and efficacy of a minimal monitoring (MINMON) strategy of delivering interferon- and ribavirin (RBV)-free, pan-genotypic direct-acting antiviral (DAA) therapy to treat active hepatitis C virus (HCV) in HCV treatment naïve participants, with or without HIV-1 co-infection, and with no evidence of decompensated cirrhosis.

The MINMON intervention included four components: 1) No pre-treatment HCV genotyping; 2) Entire 12-week treatment course (84 tablets) dispensed to participants at study entry; 3) No scheduled on-treatment laboratory monitoring or clinic visits prior to SVR evaluation scheduled 24 weeks following entry; 4) Remote contact with participants at week 4 for adherence counseling and locator update, and week 22 for scheduling of SVR visit and locator update.

At study entry, all participants received a single-tablet, fixed-dose combination (FDC) of sofosbuvir/velpatasvir (SOF/VEL) for 12 weeks.

The trial was designed to accrue 400 adult participants who may be co-infected with HIV-1 (limited to no more than 200 participants), and whose liver disease state is either no cirrhosis (defined by Fibrosis-4 score) or compensated cirrhosis (defined by Fibrosis-4 and Child-Turcotte-Pugh (CTP) scores, and limited to no more than 80 participants). Accrual from research sites in the United States was limited to no more than 132 participants.

The study proceeded in two steps: Step 1: MINMON intervention and Step 2: post-MINMON follow up.

During Step 1 (MINMON intervention), participants were contacted remotely at week 4 to inquire about study medication adherence and confirm locator information, and again at week 22 to schedule the sustained virologic response (SVR) evaluation and confirm locator information. Unplanned in-person clinic visits before week 22 were permissible to address common treatment toxicities that could not be managed remotely. The primary efficacy outcome measure, sustained virologic response (SVR), was evaluated starting at the week 24 study visit. Early discontinuation of treatment did not alter the timing of the SVR evaluation. If the week 24 visit was missed, SVR could be evaluated at any time up to 76 weeks following study entry.

Following SVR evaluation, participants entered Step 2 for two additional post-SVR evaluation study visits at weeks 48 and 72. Participants were contacted remotely at weeks 42 and 68 to schedule such visits. The schedule of additional post-MINMON evaluation visits were dependent on the week of Step 2 entry.

In version 1 of the study, total study duration was up to 76 weeks. Due to the COVID-19 Pandemic, the window of the week 72 visit was extended for participants who completed SVR evaluations and registered to Step 2 to October 31, 2020 for US sites and to February 28, 2021 for non-US sites. This extension did not alter the window for SVR evaluation.

All scheduled in-clinic study visits included a physical exam, blood collection, and collection of plasma samples. For participants able to become pregnant, pregnancy testing was conducted at screening, entry, and at any in-clinic visit during Step 1 if pregnancy was suspected. Liver Elastography was an optional evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Active Hepatitis C (HCV) infection, defined by HCV RNA >1000 international units (IU/mL) within 35 days prior to study entry
* HCV treatment naïve
* Liver disease staged as either non-cirrhotic (Fibrosis-4 (FIB-4) Score <3.25) or compensated cirrhotic (FIB-4 Score ≥3.25 and Child-Turcotte-Pugh (CTP) ≤Score 6) within 35 days prior to study entry
* HIV-1 negative, or HIV-1 positive with either a) Non-efavirenz containing antiretroviral therapy (ART) started at least 14 days prior to study entry with plasma HIV-1 RNA <400 copies/mL within 90 days prior to study entry or b) not taking ART and CD4+ cell count >350 cells/uL within 90 days prior to study entry
* The following laboratory values obtained within 35 days prior to study entry:

  * Albumin >3.0 g/L
  * Hemoglobin >8.0 g/dL for women; >9.0 g/dL for men
  * Platelet count >50,000/mm^3
  * Calculated creatinine clearance (CrCl) >30 mL/min
  * Aspartate aminotransferase (AST) <10 times the upper limit of the normal range (ULN)
  * Alanine transaminase (ALT) <10 times the ULN
  * Total bilirubin <1.5 times the ULN for participants not on atazanavir (ATV); <3 times the ULN for participants on ATV
  * International normalized ratio (INR) <1.5 times the ULN
* For females of reproductive potential, a negative serum or urine pregnancy test within 48 hours prior to study entry
* All participants of reproductive potential must have agreed not to participate in conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization) while on study treatment and for 6 weeks after stopping study treatment
* If participating in sexual activity that could lead to pregnancy, the all participants of reproductive potential had to agree to use at least one reliable methods of contraception while on study treatment and for 6 weeks after stopping study treatment
* Participants who were not of reproductive potential were eligible without requiring the use of contraceptives.
* Life expectancy >12 months
* Ability and willingness to be contacted remotely
* Ability and willingness of participant to provide informed consent.

Exclusion Criteria:

* Positive for hepatitis B virus (HBV) surface antigen
* For cirrhotic participants, CTP score >6 corresponding to Class B or C
* Breastfeeding or pregnancy
* Known allergy/sensitivity or any hypersensitivity to components of study drugs or their formulation
* Active drug or alcohol use or dependence and other conditions that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Acute or serious illness requiring systemic treatment and/or hospitalization within 35 days prior to study entry
* For HIV positive participants, presence of active or acute AIDS-defining opportunistic infections within 35 days prior to study entry
* Any history of hepatic decompensation including ascites, spontaneous bacterial peritonitis, hepatic encephalopathy, hepatorenal syndrome, and/or bleeding esophageal varices
* Use of prohibited medications within the past 14 days prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2021-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Solomon, MBBS, PhD, MPH, Study Chair — Johns Hopkins University
Locations (38):
- United States (30):
  - Alabama CRS (31788), Birmingham, Alabama
  - University of Southern California (1201), Los Angeles, California
  - UCLA CARE Center CRS (601), Los Angeles, California
  - Ucsd, Avrc Crs (701), San Diego, California
  - Ucsf Aids Crs (801), San Francisco, California
  - University of Colorado Hospital CRS (6101), Aurora, Colorado
  - Whitman Walker Health CRS (31791), Washington D.C., District of Columbia
  - The Ponce de Leon Center CRS (5802), Atlanta, Georgia
  - Northwestern University CRS (2701), Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS (2702), Chicago, Illinois
  - Johns Hopkins University CRS (201), Baltimore, Maryland
  - Massachusetts General Hospital (MGH) CRS (101), Boston, Massachusetts
  - Brigham and Women's Hosp. ACTG CRS (107), Boston, Massachusetts
  - Washington U CRS (2101), St Louis, Missouri
  - New Jersey Medical School Clinical Research Center CRS (31786), Newark, New Jersey
  - Weill Cornell Chelsea CRS (7804), New York, New York
  - Columbia Physicians and Surgeons CRS (30329), New York, New York
  - Weill Cornell Upton CRS (7803), New York, New York
  - University of Rochester Adult HIV Therapeutic Strategies Network CRS (31787), Rochester, New York
  - Unc Aids Crs (3201), Chapel Hill, North Carolina
  - Greensboro CRS (3203), Greensboro, North Carolina
  - Univ. of Cincinnati CRS (2401), Cincinnati, Ohio
  - Case CRS (2501), Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS (2301), Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS (6201), Philadelphia, Pennsylvania
  - Pittsburgh CRS (1001), Pittsburgh, Pennsylvania
  - The Miriam Hospital ACTG CRS (2951), Providence, Rhode Island
  - Vanderbilt Therapeutics (VT) CRS (3652), Nashville, Tennessee
  - Trinity Health and Wellness Center CRS (31443), Dallas, Texas
  - Houston AIDS Research Team CRS (31473), Houston, Texas
- Brazil (2):
  - Hospital Nossa Senhora da Conceicao CRS (12201), Porto Alegre, Rio Grande do Sul
  - Instituto de Pesquisa Clinica Evandro Chagas (12101), Rio de Janeiro
- Puerto Rico-AIDS CRS (5401), San Juan, Puerto Rico
- South Africa (2):
  - University of the Witwatersrand Helen Joseph (WITS HJH) CRS (11101), Johannesburg, Gauteng
  - Family Clinical Research Unit (FAM-CUR) CRS (8950), Cape Town, West Cape
- Thailand (2):
  - Thai Red Cross AIDS Research Centre (TRC-ARC) CRS (31802), Bangkok, Patumwan
  - Chiang Mai University HIV Treatment CRS (31784), Chiang Mai
- Joint Clinical Research Centre (JCRC) (12401), Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Torres TS, Saha PT, Smeaton L, Wimbish C, Kliemann DA, Avihingsanon A, Kityo C, Bennet JA, Van Schalkwyk M, Linas B, Nunes EP, Robbins GK, Wyles D, Naggie S, Sulkowski M, Cardoso SW, Solomon S. Impact of a minimal monitoring HCV treatment approach on Health-Related Quality of Life. Qual Life Res. 2025 Jun;34(6):1683-1694. doi: 10.1007/s11136-025-03922-1. Epub 2025 Feb 28. PMID 40019678
- [Derived] Han WM, Solomon SS, Smeaton L, Avihingsanon A, Wagner Cardoso S, Li J, Parvangada A, Sulkowski M, Naggie S, Martin R, Mo H, Maiorova E, Wyles D. Reinfection and Resistance Associated Substitutions Following a Minimal Monitoring Approach for Hepatitis C Virus Treatment in MINMON Trial. Clin Infect Dis. 2025 Jul 18;80(6):1293-1301. doi: 10.1093/cid/ciae627. PMID 39702964
- [Derived] Sowah LA, Smeaton L, Brates I, Bhattacharya D, Linas B, Kreter B, Wagner-Cardoso S, Solomon S, Sulkowski M, Robbins GK. Perspectives on Adherence From the ACTG 5360 MINMON Trial: A Minimum Monitoring Approach With 12 Weeks of Sofosbuvir/Velpatasvir in Chronic Hepatitis C Treatment. Clin Infect Dis. 2023 Jun 8;76(11):1959-1968. doi: 10.1093/cid/ciad034. PMID 36694361
- [Derived] Solomon SS, Wagner-Cardoso S, Smeaton L, Sowah LA, Wimbish C, Robbins G, Brates I, Scello C, Son A, Avihingsanon A, Linas B, Anthony D, Nunes EP, Kliemann DA, Supparatpinyo K, Kityo C, Tebas P, Bennet JA, Santana-Bagur J, Benson CA, Van Schalkwyk M, Cheinquer N, Naggie S, Wyles D, Sulkowski M. A minimal monitoring approach for the treatment of hepatitis C virus infection (ACTG A5360 [MINMON]): a phase 4, open-label, single-arm trial. Lancet Gastroenterol Hepatol. 2022 Apr;7(4):307-317. doi: 10.1016/S2468-1253(21)00397-6. Epub 2022 Jan 10. PMID 35026142
- See also: DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1 — http://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — http://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids
- See also: NIH. BLAST® Basic Local Alignment Search Tool. US National Library of Medicine, National Center for Biotechnology Information, NIH; 2021 — http://blast.ncbi.nlm.nih.gov/Blast.cgi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from October 2018 to July 2019 at 38 sites in Brazil, South Africa, Thailand, Uganda, and the United States.
Pre-assignment Details: There was no randomization in this study. Enrollment from sites located in the United States was restricted to 132 participants. Enrollment of participants having compensated cirrhosis was limited to no more than 80 participants, and enrollment of people living with HIV was limited to no more than 200 participants.
Groups:
- MINMON 24 Weeks With SOF/VEL 12 Weeks: Participants received Sofosbuvir/Velpatasvir (SOF/VEL [Tradename: Epclusa®]) tablet for 12 weeks with a minimal monitoring (MINMON) strategy for 24 weeks
  Sofosbuvir/Velpatasvir (SOF/VEL): 400/100 mg fixed-dose combination (FDC) tablet administered orally once daily with or without food.
  Minimal Monitoring (MINMON) Strategy: MINMON Strategy:
  1. No pre-treatment HCV genotyping
  2. Entire treatment course (84) tablets of SOF/VEL administered to participants at study entry
  3. No scheduled on-treatment laboratory monitoring or clinic visits
  4. Remote contact with participants at week 4 and week 22
Period: Step 1: MINMON Intervention
Arm/Group | MINMON 24 Weeks With SOF/VEL 12 Weeks
Started | 400
Completed | 396
Not Completed | 4
Not completed — Lost to Follow-up | 3
Not completed — Protocol Violation | 1
Period: Step 2:Post-MINMON
Arm/Group | MINMON 24 Weeks With SOF/VEL 12 Weeks
Started | 396
Completed | 362
Not Completed | 34
Not completed — Death | 2
Not completed — Lost to Follow-up | 30
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Participants who enrolled into study and received first dose of study medication.
Arm/Group | MINMON 24 Weeks With SOF/VEL 12 Weeks
Number analyzed (Participants) | 399
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47 [37 to 57]
Age, Customized [Count of Participants; unit: Participants]
  20 to 29 years | 33
  30 to 39 years | 95
  40 to 49 years | 100
  50 to 59 years | 97
  60 to 69 years | 55
  70 to 79 years | 18
  80+ years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139
  Male | 260
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 95
  Not Hispanic or Latino | 289
  Unknown or Not Reported | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 113
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 72
  White | 166
  More than one race | 0
  Unknown or Not Reported | 47
Region of Enrollment [Number; unit: participants]
  Brazil | 131
  South Africa | 12
  Thailand | 110
  Uganda | 15
  United States | 131
Gender Identity [Count of Participants; unit: Participants] — Persons identifying across the transgender spectrum includes endorsement of any gender identities that do not match sex assigned at birth including transgender, genderqueer, gender variant or gender non-conforming, and other gender self-identities.
  Participants
    Cisgender | 377
    Transgender Spectrum | 22
HIV-infection Status [Count of Participants; unit: Participants]
  HIV-1 infection absent | 233
  HIV-1 infection present | 166
Cirrhosis Status [Count of Participants; unit: Participants] — Cirrhosis present defined as Fibrosis-4 (FIB-4) Score >= 3.25 and cirrhosis absent is defined as FIB-4 Score <3.25
  Participants
    Cirrhosis present | 34
    Cirrhosis absent | 365
HCV RNA [Median (Inter-Quartile Range); unit: Log10 IU/ml] | 6.1 [5.6 to 6.6]
HCV Genotype [Count of Participants; unit: Participants] — Genotypes determined via Sanger sequencing of a short (~325 base pair) fragment sequence of the NS5B region and phylogenetic determination of genotype using Basic Local Alignment Search Tool (NIH BLAST; 2021). Specimen from 3 participants did not provide results and are listed as 'Unknown Genotype'.
  Participants
    Genotype 1 | 249
    Genotype 2 | 26
    Genotype 3 | 80
    Genotype 4 | 26
    Genotype 5 | 3
    Genotype 6 | 11
    Genotype 7 | 1
    Unknown Genotype | 3
Self Reported History of Substance Use [Count of Participants; unit: Participants] — History of substance use is defined as any current or previous usage of any of the following on the WHO ASSIST questionnaire at study entry: amphetamines, hallucinogens, cocaine, opioids, or sedatives. Current use is defined as use at least once in the past three months prior to study entry.
  Participants
    Currently | 56
    Previously | 170
    Never | 171
    Not evaluated | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 (SVR12)
Description: SVR12 was defined as plasma HCV RNA less than the lower limit of quantification (LLOQ) from the earliest sample drawn at least 22 weeks following study treatment initiation (i.e. at a visit scheduled at least 10 weeks after scheduled end of study treatment). Participants without any HCV RNA result at least 22 weeks after treatment initiation will be considered as having HCV RNA greater than the LLOQ.
  LLOQ was defined as <15 IU/mL for results tested at USA centralized testing laboratory Quest using the "Roche COBAS® HCV Quantitative nucleic acid test for use on the COBAS® 6800/8800" assays for quantitation (and detection) of HCV, and <12 IU/mL for results tested at regional international labs using "Abbott RealTime HCV" assay for quantitation (and detection) of HCV.
  A two-sided 95%, confidence interval was calculated for this percentage using the Wilson (score) method.
Time Frame: From at least 22 weeks and up to 76 weeks from treatment initiation
Population: Participants who enrolled and received first dose of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MINMON 24 Weeks With SOF/VEL 12 Weeks
Number analyzed (Participants) | 399
percentage of participants | 95.0 [92.4 to 96.7]

2. Primary Outcome: Percentage of Participants With an Occurrence of Serious Adverse Events According to International Council for Harmonization (ICH) Criteria
Description: Serious adverse events (SAEs) as defined by ICH guidelines.
  A two-sided, 95% confidence interval was calculated for the percentage using the Wilson (score) method.
Time Frame: From treatment initiation to 28 weeks
Population: Participants who received first dose of study medication and had at least one post-entry evaluation for adverse events.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MINMON 24 Weeks With SOF/VEL 12 Weeks
Number analyzed (Participants) | 397
percentage of participants | 3.5 [2.1 to 5.8]

3. Secondary Outcome: Percentage of Participants With at Least One Unplanned Clinic Visit Prior to SVR12 Evaluation
Description: According to the study minimal monitoring intervention, there were no planned clinic visits prior to study week 24, when SVR12 was scheduled to be evaluated. An unplanned clinic visit was defined as an in-clinic visit occurring from treatment initiation to up to week 22.
  A two-sided, 95% confidence interval was calculated for the percentage using the Wilson (score) method.
Time Frame: From treatment initiation to 22 weeks
Population: Participants who enrolled and received first dose of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MINMON 24 Weeks With SOF/VEL 12 Weeks
Number analyzed (Participants) | 399
percentage of participants | 3.8 [2.3 to 6.1]

4. Secondary Outcome: Percentage of Participants With an Occurrence of One or More Non-serious, Grade >= 3 Adverse Event (AE), or Treatment Limiting AE.
Description: AEs included all primary diagnoses, primary signs/symptoms, and primary laboratory abnormalities that either had severity grade ≥ 3 or led to a change in study medication. Serious Adverse Events (SAE) by International Council for Harmonization (ICH) criteria were excluded as they contributed to the primary safety outcome measure.
  Severity grading was based on DAIDS AE Grading Table, Corrected Version 2.1.
  A two-sided, 95% confidence interval was calculated for the percentage using the Wilson (score) method.
Time Frame: From treatment initiation to 28 weeks
Population: Participants who received first dose of study medication and had at least one post-entry evaluation for adverse events.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MINMON 24 Weeks With SOF/VEL 12 Weeks
Number analyzed (Participants) | 397
percentage of participants | 5.8 [5.1 to 6.6]

5. Secondary Outcome: Percentage of Participants Who Prematurely Discontinued HCV Study Medications
Description: Since there were no planned clinic visits during the 12 week study medication period, the last dose of study treatment was self-reported by participants, and recorded at the SVR evaluation visit at 24 weeks. Premature treatment discontinuation was defined when the self-reported final dose date was <11 weeks (<77 days) after the date of initial dose (accounting for any reported treatment holds). Participants discontinuing study follow up without information about completion of HCV study medications were counted as having prematurely discontinued medications.
  A two-sided, 95% confidence interval was calculated for the percentage using the Wilson (score) method.
Time Frame: From at least 22 weeks and up to 76 weeks from treatment initiation
Population: Participants who enrolled into study and received first dose of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MINMON 24 Weeks With SOF/VEL 12 Weeks
Number analyzed (Participants) | 399
percentage of participants | 1.0 [0.4 to 2.5]

ADVERSE EVENTS:
Time Frame: From treatment initiation to study completion at week 72. The week 72 window was extended for participants who completed SVR evaluations and registered to Step 2 to October 31, 2020 for US sites and to February 28, 2021 for non-US sites in response to COVID-19, up to a maximum of 110 weeks.
Description: For participants who received first dose of SOF/VEL and had at least one post-entry evaluation for AEs. Post-entry, all signs/symptoms, diagnoses, or abnormal laboratory findings new in onset or aggravated in severity or frequency from the baseline condition and meeting any of the following criteria were reported: ≥ Grade 3, led to change in SOF/VEL regardless of grade, or met expedited AE or ICH SAE guidelines. The DAIDS AE Grading Table (Correct V2.1) and Expedited AE Manual (V2.0) were used.
Arm/Group | MINMON 24 Weeks With SOF/VEL 12 Weeks
All-Cause Mortality (participants affected / at risk) | 2/397
Serious Adverse Events (participants affected / at risk) | 31/397
Other Adverse Events (participants affected / at risk) | 58/397
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MINMON 24 Weeks With SOF/VEL 12 Weeks (N=397)
Anaemia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Acute right ventricular failure (Cardiac disorders) | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Haemoglobin decreased (Investigations) | 2
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ischaemic stroke (Nervous system disorders) | 1
Neuromyelitis optica spectrum disorder (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1
Depression (Psychiatric disorders) | 1
Intentional self-injury (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 1
Persistent depressive disorder (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Schizoaffective disorder depressive type (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Ureterolithiasis (Renal and urinary disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Substance use (Social circumstances) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MINMON 24 Weeks With SOF/VEL 12 Weeks (N=397)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Acute left ventricular failure (Cardiac disorders) | 1
Left ventricular failure (Cardiac disorders) | 1
Gilbert's syndrome (Congenital, familial and genetic disorders) | 1
Chorioretinopathy (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 3
Blood creatinine increased (Investigations) | 5
Blood pressure increased (Investigations) | 2
Creatinine renal clearance decreased (Investigations) | 22
Haemoglobin decreased (Investigations) | 1
Weight decreased (Investigations) | 3
Abnormal loss of weight (Metabolism and nutrition disorders) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Tongue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 1
Depressive symptom (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Urine abnormality (Renal and urinary disorders) | 1
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Hypertension (Vascular disorders) | 1
Hypertensive urgency (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.

DOCUMENTS (3):
  • Study Protocol (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/10/NCT03512210/Prot_001.pdf
  • Statistical Analysis Plan (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/10/NCT03512210/SAP_002.pdf
  • Informed Consent Form (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/10/NCT03512210/ICF_000.pdf